CLINICAL TRIAL: NCT00203723
Title: A Comparison Study of Combined ECT and Risperidone Versus ECT Alone for Treatment Resistant Depression.
Brief Title: Use of Risperidone in ECT for Treatment Resistant Depression
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Janssen, LP (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UCLA IRB #03-10-049-01; RIS-DEP-405
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2006-05-18 (Estimated); Status verified 2006-05

CONDITIONS: Major Depression
Keywords: mood disorder; affective disorder; depression; treatment-resistant
MeSH Terms: conditions — Depressive Disorder, Major; Mood Disorders; Depression | interventions — Risperidone

INTERVENTIONS:
Drug: Risperidone

SUMMARY:
The purpose of this study is to determine if the combination of risperidone and ECT improves a patient's response in depression compared to ECT alone.

DETAILED DESCRIPTION:
Medication resistance to antidepressant therapy, or Treatment-Resistant Depression (TRD), is the main reason, if not main indication, for which patients are presently referred for electroconvulsive therapy (ECT) in hopes of a rapid, definitive response (APA 2001 ECT Task Force Report). While the causes of TRD remain unclear, this category of patients includes those who have incomplete remission, those who relapse rapidly and frequently, those who have psychotic depression, those who develop chronic depression, and those who often have comorbid medical and psychiatric illness (Sackeim 2001, Sharma 2001, Fava and Davidson 1996, Thase 1995). Moreover, while increased age per se is not a barrier to antidepressant response, many elderly, especially those with comorbid medical or neurological illness, are unable to tolerate courses of aggressive pharmacotherapy or seem to have a less robust response to pharmacotherapy, and possibly to ECT alone, with significant residual functional and cognitive impairment (Reynolds 1998, Stoudemire 1998, Lebowitz 1997, Gurland 1991).

Compared to patients who are not medication resistant, who generally retain the highest likelihood of response to ECT alone, patients with TRD have a lower response rate to ECT with average estimates of response to ECT alone between 50-60% (APA 2001 ECT Task Force). Additionally, while ECT for most patients may provide acute remission, those patients with TRD remain at high risk for rapid relapse (Sackeim 2001, Petrides 2001, Sackeim 1990, Aronson 1987). Consequently, ECT alone may be insufficient to achieve remission or to prevent relapse. Interestingly, resistance to some types of medication was found also to predict resistance to ECT alone, i.e., resistance to tricyclic antidepressants correlated with a less likely response to ECT, though the same prediction did not hold for serotonin reuptake inhibitors (Prudic 1996, Prudic 1990).

In general, for some patients with TRD, studies support the use of combined medication approaches, and specifically, have demonstrated the safety, tolerability and effectiveness of an antidepressant with an antipsychotic medication, though usually for patients with comorbid psychosis (Wheeler 2000, Shelton 1999, Barak 1999). Case reports exist in the ECT literature about the safety and tolerability of ECT and antipsychotics, and improved efficacy, albeit generally for patients with psychotic depression or other treatment resistant psychoses (Kupchik 2000, Bhatia 1998, Ranjan 1996, Farah, Beale, and Kellner 1995, Minter 1979). However, no studies systematically, or prospectively, investigate whether the specific combination of ECT plus an atypical antipsychotic offers a true treatment alternative to improved efficacy of ECT for patients with TRD.

This study reviews the experience and outcome of combining ECT and an atypical antipsychotic medication, risperidone, for TRD in various populations in an academic, university-based setting, and furthermore, explores in a pilot randomized open-label study whether ECT plus risperidone bears closer scrutiny in more rigorous study designs as a novel treatment approach.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 to 89 years, inclusive
* Male or female
* Inpatient or outpatient ECT with a current diagnosis of unipolar or bipolar depression, with or without psychosis, according to DSM-IV criteria. HAM-D (17-item) score > 17 and MADRS score > 18 at screening and at first treatment session.

Exclusion Criteria:

* MMSE < 23
* Inability to consent to ECT
* Current diagnosis of schizophrenia or schizoaffective disorder
* Current diagnosis of Parkinson's Disease or any Dementia, including Lewy Body Disease
* History of allergic reaction to risperidone
* History of Neuroleptic Malignant Syndrome
* Current pregnancy or positive urine pregnancy test
* Women who are breast-feeding
* Active alcohol or illicit substance abuse

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45
Dates: Start 2005-03; Study Completion 2006-05

PRIMARY OUTCOMES:
Scores on depression scales after 6 ECT treatments

SECONDARY OUTCOMES:
Scores on Clinical Global Impression Scales and Symptom Checklist

CONTACTS AND LOCATIONS:
Overall Officials: Randall Espinoza, MD, MPH, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Npi&H, Los Angeles, California, United States